CLINICAL TRIAL: NCT00152386
Title: A Phase III Multicentre, Double Blind, Placebo-controlled, Parallel Group 52-week Study to Assess the Efficacy and Safety of 2 Dose Regimens of Lyophilised CDP870 as Additional Medication to Methotrexate in the Treatment of Signs and Symptoms and Preventing Structural Damage in Patients With Active Rheumatoid Arthritis Who Have an Incomplete Response to Methotrexate
Brief Title: A Placebo Controlled Study to Assess Efficacy and Safety of Certolizumab Pegol in the Treatment of Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C87027; 2004-002993-49 (EudraCT Number)
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis, CDP870; Certolizumab pegol, Cimzia
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Certolizumab Pegol

INTERVENTIONS:
Drug: Certolizumab pegol (CDP870)

SUMMARY:
Patients will be assigned to one of three treatment groups. Study medication is administered over a 52 week study duration.

ELIGIBILITY:
Inclusion Criteria:

* Male and female, aged at least 18 years old at the Screening visit.
* A clear chest X-ray within 3 months prior to Baseline visit.
* A diagnosis of adult-onset RA (of at least six months duration but not longer than 15 years prior to Screening) as defined by the 1987 American College of Rheumatology classification criteria.
* Active RA disease at Screening and Baseline as defined by:

  * ≥9 tender joints.
  * ≥9 swollen joints. and fulfilling 1 of the following 2 criteria:
  * ≥30 mm/hour ESR (Westergren), or
  * CRP >15 mg/L.
* Must have received a stable dose of MTX with or without folic acid for at least 3 months prior to Baseline visit. The minimum dose is 10 mg MTX weekly.
* Patient must be willing to attend for a Week 52 X-ray of the hands and feet even if they are no longer receiving study treatment but have not withdrawn their informed consent.

Exclusion Criteria:

* A diagnosis of any other inflammatory arthritis e.g., psoriatic arthritis or ankylosing spondylitis.
* A secondary, non-inflammatory type of arthritis (e.g. OA or fibromyalgia) that in the Investigator's opinion is symptomatic enough to interfere with evaluation of the effect of CDP870 on the patient's primary diagnosis of RA.
* A history of an infected joint prosthesis at any time with prosthesis still in situ.
* Does not meet exclusionary concomitant medication criteria.
* A history of a lymphoproliferative disorder including lymphoma or signs and symptoms suggestive of lymphoproliferative disease at any time.
* Patients at a high risk of infection in the Investigator's opinion (e.g. leg ulcers, indwelling urinary catheter and persistent or recurrent chest infections).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 950
Dates: Start 2005-02; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of CDP870 in combination with Methotrexate in the treatment of Rheumatoid Arthritis and prevention of structural damage by measuring the ACR20 response at week 24 and change from Baseline

SECONDARY OUTCOMES:
Change from Baseline in mTSS at week 24, Change from Baseline in HAQ-DI at weeks 24 and 52, ACR20 responder rate at week 52, ACR50 and ACR70 responder rate at weeks 24 and 52

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma
Locations (76):
- United States (26):
  - Huntsville, Alabama
  - Paradise Valley, Arizona
  - La Jolla, California
  - San Diego, California
  - Denver, Colorado
  - Danbury, Connecticut
  - Washington D.C., District of Columbia
  - Aventura, Florida
  - Ocala, Florida
  - Orlando, Florida
  - Sarasota, Florida
  - Tampa, Florida
  - Coeur d'Alene, Idaho
  - Springfield, Illinois
  - Wichita, Kansas
  - Wheaton, Maryland
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Charlotte, North Carolina
  - Cleveland, Ohio
  - Dayton, Ohio
  - Duncansville, Pennsylvania
  - Charleston, South Carolina
  - Austin, Texas
  - Dallas, Texas
  - San Antonio, Texas
- Argentina (2):
  - Capital Federal
  - Córdoba
- Australia (8):
  - Camperdown
  - Coffs Harbour
  - Cotton Tree
  - Malvern
  - Shenton Park
  - Victoria Park
  - Westmead
  - Wooloongabba
- Belgium (5):
  - Antwerp
  - Brussels
  - Liège
  - Merksem
  - Sijsele
- Bulgaria (4):
  - Pleven
  - Sofia
  - Stara Zagora
  - Varna
- Canada (11):
  - Courtice
  - Hamilton
  - Kitchener
  - London
  - Mississauga
  - Montreal
  - Newmarket
  - Point Claire
  - Sainte-Foy
  - Toronto
  - Winnipeg
- Chile (4):
  - Valdivia, Las Condes
  - Santiago, Santiago Centro
  - Santiago
  - Temuco
- Rijeka, Croatia
- Czechia (7):
  - Brno
  - Brno-Bohunice
  - Ostrava Trebovice
  - Pilsen
  - Prague
  - Uherské Hradiště
  - Zlín
- Israel (4):
  - Afula
  - Haifa
  - Ramat Gan
  - Tel Aviv
- Riga, Latvia
- Russia (2):
  - Moscow
  - Saint Petersburg
- Ivano-Frankivsk, Ukraine

REFERENCES:
- [Result] Keystone E, Heijde Dv, Mason D Jr, Landewe R, Vollenhoven RV, Combe B, Emery P, Strand V, Mease P, Desai C, Pavelka K. Certolizumab pegol plus methotrexate is significantly more effective than placebo plus methotrexate in active rheumatoid arthritis: findings of a fifty-two-week, phase III, multicenter, randomized, double-blind, placebo-controlled, parallel-group study. Arthritis Rheum. 2008 Nov;58(11):3319-29. doi: 10.1002/art.23964. PMID 18975346
- [Result] van Vollenhoven RF, Felson D, Strand V, Weinblatt ME, Luijtens K, Keystone EC. American College of Rheumatology hybrid analysis of certolizumab pegol plus methotrexate in patients with active rheumatoid arthritis: data from a 52-week phase III trial. Arthritis Care Res (Hoboken). 2011 Jan;63(1):128-34. doi: 10.1002/acr.20331. PMID 20799264
- [Result] Hazes JM, Taylor P, Strand V, Purcaru O, Coteur G, Mease P. Physical function improvements and relief from fatigue and pain are associated with increased productivity at work and at home in rheumatoid arthritis patients treated with certolizumab pegol. Rheumatology (Oxford). 2010 Oct;49(10):1900-10. doi: 10.1093/rheumatology/keq109. Epub 2010 Jun 14. PMID 20547658
- [Result] Pincus T, Furer V, Keystone E, Yazici Y, Bergman MJ, Luijtens K. RAPID3 (Routine Assessment of Patient Index Data 3) severity categories and response criteria: Similar results to DAS28 (Disease Activity Score) and CDAI (Clinical Disease Activity Index) in the RAPID 1 (Rheumatoid Arthritis Prevention of Structural Damage) clinical trial of certolizumab pegol. Arthritis Care Res (Hoboken). 2011 Aug;63(8):1142-9. doi: 10.1002/acr.20481. PMID 21485024
- [Result] Curtis JR, Chen L, Luijtens K, Navarro-Millan I, Goel N, Gervitz L, Weinblatt M. Dose escalation of certolizumab pegol from 200 mg to 400 mg every other week provides no additional efficacy in rheumatoid arthritis: an analysis of individual patient-level data. Arthritis Rheum. 2011 Aug;63(8):2203-8. doi: 10.1002/art.30387. PMID 21484766
- [Result] Keystone EC, Curtis JR, Fleischmann RM, Furst DE, Khanna D, Smolen JS, Mease PJ, Schiff MH, Coteur G, Davies O, Combe B. Rapid improvement in the signs and symptoms of rheumatoid arthritis following certolizumab pegol treatment predicts better longterm outcomes: post-hoc analysis of a randomized controlled trial. J Rheumatol. 2011 Jun;38(6):990-6. doi: 10.3899/jrheum.100935. Epub 2011 Mar 1. PMID 21362764
- [Result] Curtis JR, Luijtens K, Kavanaugh A. Predicting future response to certolizumab pegol in rheumatoid arthritis patients: features at 12 weeks associated with low disease activity at 1 year. Arthritis Care Res (Hoboken). 2012 May;64(5):658-67. doi: 10.1002/acr.21600. PMID 22231904
- [Result] Paul S, Marotte H, Kavanaugh A, Goupille P, Kvien TK, de Longueville M, Mulleman D, Sandborn WJ, Vande Casteele N. Exposure-Response Relationship of Certolizumab Pegol and Achievement of Low Disease Activity and Remission in Patients With Rheumatoid Arthritis. Clin Transl Sci. 2020 Jul;13(4):743-751. doi: 10.1111/cts.12760. Epub 2020 Apr 1. PMID 32100960
- [Derived] Curtis JR, Winthrop K, O'Brien C, Ndlovu MN, de Longueville M, Haraoui B. Use of a baseline risk score to identify the risk of serious infectious events in patients with rheumatoid arthritis during certolizumab pegol treatment. Arthritis Res Ther. 2017 Dec 15;19(1):276. doi: 10.1186/s13075-017-1466-y. PMID 29246162
- [Derived] Combe B, Furst DE, Keystone EC, van der Heijde D, Luijtens K, Ionescu L, Goel N, Emery P. Certolizumab Pegol Efficacy Across Methotrexate Regimens: A Pre-Specified Analysis of Two Phase III Trials. Arthritis Care Res (Hoboken). 2016 Mar;68(3):299-307. doi: 10.1002/acr.22676. PMID 26238672
- [Derived] van der Heijde D, Keystone EC, Curtis JR, Landewe RB, Schiff MH, Khanna D, Kvien TK, Ionescu L, Gervitz LM, Davies OR, Luijtens K, Furst DE. Timing and magnitude of initial change in disease activity score 28 predicts the likelihood of achieving low disease activity at 1 year in rheumatoid arthritis patients treated with certolizumab pegol: a post-hoc analysis of the RAPID 1 trial. J Rheumatol. 2012 Jul;39(7):1326-33. doi: 10.3899/jrheum.111171. Epub 2012 May 15. PMID 22589265
- [Derived] Strand V, Mease P, Burmester GR, Nikai E, Coteur G, van Vollenhoven R, Combe B, Keystone EC, Kavanaugh A. Rapid and sustained improvements in health-related quality of life, fatigue, and other patient-reported outcomes in rheumatoid arthritis patients treated with certolizumab pegol plus methotrexate over 1 year: results from the RAPID 1 randomized controlled trial. Arthritis Res Ther. 2009;11(6):R170. doi: 10.1186/ar2859. Epub 2009 Nov 12. PMID 19909548
- [Derived] Kavanaugh A, Smolen JS, Emery P, Purcaru O, Keystone E, Richard L, Strand V, van Vollenhoven RF. Effect of certolizumab pegol with methotrexate on home and work place productivity and social activities in patients with active rheumatoid arthritis. Arthritis Rheum. 2009 Nov 15;61(11):1592-600. doi: 10.1002/art.24828. PMID 19877104